CLINICAL TRIAL: NCT04134429
Title: Continuous Monitoring of Health Data With a Wearable Device in Pediatric Patients Undergoing Chemotherapy for Cancer - a Feasibility Pilot Study
Brief Title: Feasibility of Monitoring Health Data in Pediatric Patients Undergoing Chemotherapy
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Bern 2019 WD Pilot
Record Dates: First submitted 2019-09-12; First posted 2019-10-22 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Cancer; Febrile Neutropenia; Chemotherapy-induced Neutropenia; Oncology
Keywords: wearable device; Everion®; Fever and Neutropenia; Pediatric Oncology
MeSH Terms: conditions — Neoplasms; Febrile Neutropenia; Fever; Neutropenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Everion®: The Everion® will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear it all the time, with exception of the time needed for battery charging and the patients' hygiene.
  Interventions: Device: Everion

INTERVENTIONS:
Device: Everion — The Everion® device, by Biovotion, Zurich, is a on-skin wearable device measuring health data.

SUMMARY:
In this pilot study the feasibility of continous monitoring of health data with a small, on-skin wearable device (the Everion®, by Biovotion, Zurich) in pediatric patients under chemotherapy for cancer, is studied. Feasibility is assessed by the number of patients wearing the device on seven consecutive days for at least 18h/day, what will be measured by monitored heart rate. Study duration for each participant is 14 days.

DETAILED DESCRIPTION:
No study has proved feasibility of continuous monitoring of health data with a small wearable device such as the device Everion® in pediatric patients. It is not known if children tolerate the device and if data quality sustains with smaller arm circumferences or when worn on the upper leg. Neither is it known if parents and/or patients can and are willing to handle the device in ambulant setting. Therefore, this pilot study assesses the feasibility of continous monitoring of health data with a small, on-skin wearable device (the Everion®, by Biovotion, Zurich) in pediatric patients under chemotherapy for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy treatment because of any malignancy, expected to last ≥1 months at time of recruitment for myelosuppressive therapy or at least one cycle of myeloablative therapy.
* Age 1 month to <18 years at time of recruitment
* Written informed consent from patients and/or parents

Exclusion Criteria:

* Local skin diseases prohibiting wearing of the device.
* Denied written informed consent from patients and/or parent

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients under chemotherapy for any malignancy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Brack, MD-PhD, Principal Investigator — Pediatric Hematology/Oncology, Inselspital, Bern University Hospital; Christa Koenig, MD, Study Chair — Pediatric Hematology/Oncology, Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The coded study data (from the WD and clinical data) will be uploaded to figshare and made publically available for other researchers.
Time Frame: After publication of the study results.
Access Criteria: Open access

REFERENCES:
- [Result] Koenig C, Ammann RA, Kuehni CE, Roessler J, Brack E. Continuous recording of vital signs with a wearable device in pediatric patients undergoing chemotherapy for cancer-an operational feasibility study. Support Care Cancer. 2021 Sep;29(9):5283-5292. doi: 10.1007/s00520-021-06099-8. Epub 2021 Mar 3. PMID 33655413

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Everion®
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everion®
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 6 [2 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 20
Type of malignancy [Count of Participants; unit: Participants]
  Acute lymphoblastic leukemia | 12
  Other hematologic malignancies | 2
  Central nervous system tumor | 3
  Solid tumor | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Continous Monitoring of Heart Rate With the Wearable Device (WD)
Description: The primary outcome is defined as at least acceptable (≥50) quality score (worst quality 0, best quality 100) of heart rate during a cumulative duration of ≥18/24h per day (noon to noon), during ≥7 consecutive days within the 14 days of study duration (binary outcome, measured once).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Everion®
Number analyzed (Participants) | 20
Participants | 6

2. Secondary Outcome: Continous Monitoring of Oxygen Saturation With the WD
Description: At least acceptable (≥50) quality score (worst quality 0, best quality 100) of oxygen saturation during a cumulative duration of ≥18/24h per day (noon to noon), during ≥7 consecutive days within the 14 days of study duration (binary outcome, measured once).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Everion®
Number analyzed (Participants) | 20
Participants | 0

3. Secondary Outcome: Continous Monitoring of Respiration Rate With the WD
Description: At least acceptable(≥50) quality score (worst quality 0, best quality 100) of respiration rate during a cumulative duration of ≥18/24h per day (noon to noon), during ≥7 consecutive days within the 14 days of study duration (binary outcome, measured once).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Everion®
Number analyzed (Participants) | 20
Participants | 4

4. Secondary Outcome: Continous Monitoring of Core Temperature With the WD
Description: At least acceptable(≥50) quality score (worst quality 0, best quality 100) of core temperature during a cumulative duration of ≥18/24h per day (noon to noon), during ≥7 consecutive days within the 14 days of study duration (binary outcome, measured once).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Everion®
Number analyzed (Participants) | 20
Participants | 6

5. Secondary Outcome: Continous Monitoring of Heart Rate Variability With the WD
Description: At least acceptable (≥50) quality score (worst quality 0, best quality 100) of heart rate variability during a cumulative duration of ≥18/24h per day (noon to noon), during ≥7 consecutive days within the 14 days of study duration (binary outcome, measured once).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Everion®
Number analyzed (Participants) | 20
Participants | 1

6. Secondary Outcome: Continous Monitoring of Perfusion Index With the WD
Description: At least acceptable (≥50) quality score (worst quality 0, best quality 100) of perfusion index during a cumulative duration of ≥18/24h per day (noon to noon), during ≥7 consecutive days within the 14 days of study duration (binary outcome, measured once).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Everion®
Number analyzed (Participants) | 20
Participants | 6

7. Secondary Outcome: Cumulative Time of Monitoring Heart Rate With the WD
Description: Cumulative length of time with monitored heart rate with at least acceptable quality score (≥50, worst quality 0, best quality 100) per study day (continuous outcomes, measured daily).
Time Frame: 14 days
Measure: Count of Units; unit: hours
Units Other Than Participants: hours
Arm/Group | Everion®
Number analyzed (Participants) | 20
Number analyzed (hours) | 6576
hours | 3992

8. Secondary Outcome: Cumulative Time of Monitoring Oxygen Saturation With the WD
Description: Cumulative length of time with monitored oxygen saturation with at least acceptable quality score (≥50 worst quality 0, best quality 100) per study day (continuous outcomes, measured daily).
Time Frame: 14 days
Measure: Count of Units; unit: hours
Units Other Than Participants: hours
Arm/Group | Everion®
Number analyzed (Participants) | 20
Number analyzed (hours) | 6576
hours | 1103

9. Secondary Outcome: Cumulative Time of Monitoring Respiration Rate With the WD
Description: Cumulative length of time with monitored respiration rate with at least acceptable quality score (≥50, worst quality 0, best quality 100) per study day (continuous outcomes, measured daily).
Time Frame: 14 days
Measure: Count of Units; unit: hours
Units Other Than Participants: hours
Arm/Group | Everion®
Number analyzed (Participants) | 20
Number analyzed (hours) | 6576
hours | 4058

10. Secondary Outcome: Cumulative Time of Monitoring Core Temperature With the WD
Description: Cumulative length of time with monitored core temperature with at least acceptable quality score (≥50, worst quality 0, best quality 100)) per study day (continuous outcomes, measured daily).
Time Frame: 14 days
Measure: Count of Units; unit: hours
Units Other Than Participants: hours
Arm/Group | Everion®
Number analyzed (Participants) | 20
Number analyzed (hours) | 6576
hours | 4037

11. Secondary Outcome: Cumulative Time of Monitoring Heart Rate Variability With the WD
Description: Cumulative length of time with monitored heart rate variability with at least acceptable quality score (≥50, worst quality 0, best quality 100) per study day (continuous outcomes, measured daily).
Time Frame: 14 days
Measure: Count of Units; unit: hours
Units Other Than Participants: hours
Arm/Group | Everion®
Number analyzed (Participants) | 20
Number analyzed (hours) | 6576
hours | 3142

12. Secondary Outcome: Cumulative Time of Monitoring Perfusion Index With the WD
Description: Cumulative length of time with monitored perfusion index with at least acceptable quality score (≥50, worst quality 0, best quality 100) per study day (continuous outcomes, measured daily).
Time Frame: 14 days
Measure: Count of Units; unit: hours
Units Other Than Participants: hours
Arm/Group | Everion®
Number analyzed (Participants) | 20
Number analyzed (hours) | 6576
hours | 3992

13. Secondary Outcome: Device Acceptance Assessed With Questionnaires
Description: Proportion of patients and parents indicating that continuous monitoring with the wearable device (WD) is acceptable per day and per entire study duration and reasons not to wear the device.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Everion®
Number analyzed (Participants) | 20
Participants | 18

14. Secondary Outcome: Number and Description of Side Effects
Description: Number and description of side effects reported by parents and patients, if applicable. Assessed with questionnaires.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Everion®
Number analyzed (Participants) | 20
Participants
  Superficial skin lesion | 1
  irritated skin | 4
  itching | 3
  sweating | 7

15. Secondary Outcome: Effort for Investigators Assessed by Number of Contacts
Description: Effort (cumulative number of contacts) for the Investigators.
Time Frame: 14 days
Measure: Number; unit: Total number of contacts
Arm/Group | Everion®
Number analyzed (Participants) | 20
Total number of contacts | 52

16. Secondary Outcome: Effort for Investigators Assessed by Duration of Contacts
Description: Effort (cumulative duration of contacts) for the Investigators.
Time Frame: 14 days
Measure: Number; unit: minutes
Arm/Group | Everion®
Number analyzed (Participants) | 20
minutes | 390

17. Secondary Outcome: Comparison
Description: Difference between discrete measurements performed for clinical routine cares of heart rate and the mean of continuously measured heart rate within +/-10min at times of the discrete measurement.
Time Frame: 14 days
Population: The analysis of differences between discrete measurements and continuously recorded aggregates of vital signs, as defined in the protocol, was found to yield massively distorted results because rapidly changing discretely measured vital signs were compared to aggregated means covering up to 20 min. We deliberately refrain from displaying these nonmeaningful results here.
Arm/Group | Everion®
Number analyzed (Participants) | 0

18. Secondary Outcome: Exploration of Patterns Within the Vital Signs Before Episodes With Fever or Infection
Description: Exploration of potential changes in or specific patterns of all collected signals and their quality scores in combination (heart rate, oxygen saturation, respiration rate, core temperature, skin temperature, heart rate variability, perfusion index, health score (0-100, higher score means better health), galvanic skin response) , within 48 hours before and after clinical diagnosis of fever (ear temperature of ≥39.0°C, or ≥38.5°C if fever is declared for clinical reasons) with or without neutropenia and microbiologically or clinically defined infections, if applicable.
Time Frame: 14 days
Population: The 4 episodes occured in 3 of these 20 patients. The other 17 patients had no episode with fever or infection.
Measure: Number; unit: Episodes
Arm/Group | Everion®
Number analyzed (Participants) | 20
Episodes
  Episodes with fever | 3
  Episodes with Infection | 1

ADVERSE EVENTS:
Time Frame: 17 days
Arm/Group | Everion®
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everion® (N=20)
Superficial skin lesion (Skin and subcutaneous tissue disorders) | 1 (20)

LIMITATIONS AND CAVEATS:
(i) The WDs were studied for only 14 days and compliance might be different during long-term use.

(ii) The small number of patients precluded an analysis of patient factors (iii) The planned comparison of discrete measurements versus continuously was not feasible because the exact second-wise time point of discrete measurements was not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT04134429/Prot_SAP_000.pdf